CLINICAL TRIAL: NCT01364298
Title: Multicenter, Randomized, Open-label, Parallel Group, Phase IV Study to Compare the Efficacy and Safety of Gabapentin/B-complex Versus Pregabalin in the Management of Diabetic Peripheral Neuropathic Pain
Brief Title: Efficacy and Safety of Gabapentin/B-complex Versus Pregabalin in Diabetic Peripheral Neuropathy Pain Management
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck S.A. de C.V., Mexico (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMR200054-603 CL028
Record Dates: First submitted 2011-05-31; First posted 2011-06-02 (Estimated); Results first posted 2014-02-06 (Estimated); Last update posted 2014-02-06 (Estimated); Status verified 2013-12

CONDITIONS: Diabetic Peripheral Neuropathic Pain
Keywords: Gabapentin/B complex; Pregabalin; Pain; Neuropathic; Gavindo; Lyrica
MeSH Terms: conditions — Pain | interventions — Pregabalin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gabapentin/B-complex (Experimental)
  Interventions: Drug: Gabapentin/B-complex
- Pregabalin (Active Comparator)
  Interventions: Drug: Pregabalin

INTERVENTIONS:
Drug: Gabapentin/B-complex — Gabapentin/B-complex (Gavindo®) tablet will be administered orally at an initial dose of 300 milligram per day (mg/day) on Day 1, followed by 600 mg/day (one 300 milligram [mg] tablet every 12-hour) on Day 2, then 900 mg/day (one 300 mg tablet every 8-hour) on Day 7, then 1800 mg/day (two 300 mg tablets every 8-hour) on Day 21, then 2700 mg/day (three 300 mg tablets every 8-hour) on Day 35, and finally 3600 mg/day (four 300 mg tablets every 8-hour) on Days 56 and 84. Maximum dose allowed will be 3600 mg/day. The total duration of treatment will be 84 days (12 weeks).
  Other Names: Gavindo®
  Arms: Gabapentin/B-complex
Drug: Pregabalin — Pregabalin (Lyrica®) capsule will be administered orally at an initial dose of 150 mg/day (one 75 mg capsule every 12-hour) from Day 1 to 7, followed by 300 mg/day (one 150 mg capsule every 12-hour) on Day 7, then 600 mg/day (two 150 mg capsule every 12-hour) on Days 21, 35, 56 and 84. Maximum dose allowed will be 600 mg/day. The total duration of treatment will be 84 days (12 weeks).
  Other Names: Lyrica®
  Arms: Pregabalin

SUMMARY:
This is a multicenter, randomized, open-label, parallel, Phase 4 clinical trial to compare efficacy and safety of gabapentin/B-complex versus pregabalin in diabetic peripheral neuropathy pain (DPNP) management.

DETAILED DESCRIPTION:
Primary Objective:

To compare the efficacy of gabapentin/B-complex versus pregabalin administered for 12 weeks in the treatment of pain in mild to moderate diabetic peripheral neuropathy (DPN) of acute or chronic presentation.

Secondary Objectives:

To determine the safety and tolerability of gabapentin/B-complex versus pregabalin administered for 12 weeks in the treatment of pain in mild to moderate DPN of acute or chronic presentation.

Subjects will be randomized in a 1:1 ratio to receive gabapentin/B-complex or pregabalin.

The duration of treatment per subject will be 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Females or males undististincally
* Age 18 to 70 years
* Signed informed consent (IC) by the subject
* Diabetes mellitus (DM) Type 1 or 2
* Pain due to sensorial or motor DPN of low to moderate intensity, greater than or equal to (>=) 1 year of evolution and less than or equal to (=<)5 years of being diagnosed
* Subjects who score >=40 millimeter (mm) in the visual analogue scale (VAS) of the McGill pain questionnaire (MPQ) at selection and Baseline visit, and who complete on a daily basis the numeric pain intensity (NPI) (at least 4 days a week) during the week previous to randomization and whose daily mean score is of at least 4, during the 7 days previous to randomization (with a wash-out period)
* Normal chest radiography
* Stable hypoglycemic treatment, at least 6 weeks before randomization
* Glycosylated hemoglobin (HbA1c) =<10 percent at selection visit
* Women must not be pregnant and must not have pregnancy plans during the period of the study duration
* Subjects not medicated or under analgesic stable medication during a minimum of 4 weeks, where no acceptable relief of pain is achieved; in the last case, with the corresponding wash-out period
* Women of childbearing age must submit a negative pregnancy test before treatment randomization and should use a contraceptive method medically accepted, during the study period

Exclusion Criteria:

* Suicide risk defined as a score of 2 or higher, in question 9 of the beck depression test
* Congestive heart failure Class III or IV of the New York Heart Association (NYHA)
* Subjects with serious or unstable coronary heart disease, hepatic, kidney, respiratory, hematological alterations, problems with peripheral vascular disease, or other medical or psychiatric conditions that can put in risk the participation of the subject in the study or that may lead to hospitalization during the study period
* Any condition that may lead to confusion of the diagnostic of painful DPN, in particular amputations -other than fingers/toes-, not diabetic neurological disorder and skin conditions that may affect sensation at the painful limbs
* Subjects with Baseline calculated creatinine clearance less than (<) 60 milliliter per minute (mL/min), Baseline leukocyte count < 2,500 per cubic millimeter (/mm^3), Baseline neutrophils count < 1,500/mm^3 or platelets < 100 * 10^3 /mm^3
* Subjects who have participated previously in some other study of pregabalin or gabapentin or gabapentin/B-complex, during 30 days previous to selection
* Subjects with encephalopathy caused by ammonia with alterations in the cycle of urea
* Subjects with uncontrolled closed-angle glaucoma
* Subject with presence of a disorder or an anticonvulsant treatment
* Breastfeeding women or during the first 3 months postpartum
* Morbid obesity (body mass index [BMI] >=40)
* Glycosylated hemoglobin (HbA1c) greater than (>) 10 percent
* Major surgery 3 months previous to randomization
* Any surgery 2 weeks previous to randomization process, or programmed during the study period should have been authorized by the Sponsor or appointed representative
* Blood donors 60 days previous to randomization
* Abuse or dependency of alcohol, narcotics, opioids or any other addictive substances, or energizing drinks
* History of hypersensitivity to the drugs in the study or drugs with similar chemical structures
* History or suspicion of lack of trust, poor cooperation of lack of compliance of medical treatments
* Subjects with arthritis, sciatic, fibromyalgia, restless leg syndrome, non-neuropathic muscle-skeletal pain or back chronic pain

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 353 (Actual)
Dates: Start 2011-04; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Research Manager, Study Director — Merck S.A de C.V, Mexiko, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (1):
- Research Site, Mexico City, Mexico

REFERENCES:
- [Derived] Mimenza Alvarado A, Aguilar Navarro S. Clinical Trial Assessing the Efficacy of Gabapentin Plus B Complex (B1/B12) versus Pregabalin for Treating Painful Diabetic Neuropathy. J Diabetes Res. 2016;2016:4078695. doi: 10.1155/2016/4078695. Epub 2016 Jan 17. PMID 26885528

RESULTS

PARTICIPANT FLOW:
Groups:
- Gabapentin/B-complex: Gabapentin/B-complex (Gavindo®) tablet administered orally at an initial dose of 300 milligram per day (mg/day) on Day 1, followed by 600 mg/day (one 300 milligram [mg] tablet every 12-hour) on Day 2, then 900 mg/day (one 300 mg tablet every 8-hour) on Day 7, then 1800 mg/day (two 300 mg tablets every 8-hour) on Day 21, then 2700 mg/day (three 300 mg tablets every 8-hour) on Day 35, and finally 3600 mg/day (four 300 mg tablets every 8-hour) on Days 56 and 84. Maximum dose allowed was 3600 mg/day. The total duration of treatment was 84 days (12 weeks).
- Pregabalin: Pregabalin (Lyrica®) capsule administered orally at an initial dose of 150 mg/day (one 75 mg capsule every 12-hour) from Day 1 to 7, followed by 300 mg/day (one 150 mg capsule every 12-hour) on Day 7, then 600 mg/day (two 150 mg capsule every 12-hour) on Days 21, 35, 56 and 84. Maximum dose allowed was 600 mg/day. The total duration of treatment was 84 days (12 weeks).
Period: Overall Study
Arm/Group | Gabapentin/B-complex | Pregabalin
Started | 176 | 177
Treated | 174 | 174
Completed | 162 | 154
Not Completed | 14 | 23
Not completed — Adverse Event | 3 | 4
Not completed — Lack of adherence to treatment | 1 | 3
Not completed — Lack of Efficacy | 1 | 0
Not completed — Lost to Follow-up | 5 | 10
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Other | 1 | 3

BASELINE CHARACTERISTICS:
Population: Safety population included all the randomized participants who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Gabapentin/B-complex | Pregabalin | Total
Number analyzed (Participants) | 174 | 174 | 348
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.2 (10.5) | 54.3 (9.4) | 53.8 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 119 | 109 | 228
  Male | 55 | 65 | 120

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Average Numeric Pain Intensity Scale (NPIS) Score at Day 84
Description: An average NPIS pain score (daily average records of the past seven days) was evaluated. Numeric pain intensity scale (NPIS) is a 11-point scale, with 0 representing no pain and 10 representing the worst possible pain. The participants were asked to mark the number that best represents the current level of pain they have experienced during the previous 24 hours. Change from baseline data has been calculated as value at baseline minus value at Day 84.
Time Frame: Baseline and Day 84 (Week 12)
Population: Per protocol population (PPP) included all the treated participants who showed no major protocol violations and were compliant with study inclusion criteria and with the proper administration of the study drug. 'n' signifies number of participants who were evaluable for specified categories at different time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Gabapentin/B-complex | Pregabalin
Number analyzed (Participants) | 147 | 123
units on a scale
  Baseline (n=147, 123) | 6.7 (1.5) | 6.8 (1.4)
  Change at Day 84 (n=146, 122) | 3.905 (2.639) | 4.260 (2.329)

2. Secondary Outcome: Change From Baseline in Leeds Assessment of Neuropathic Symptoms and Signs (LANSS) Scale Score at Day 84
Description: The LANSS scale score is 7-item pain scale that consists of grouped sensory description and sensory examination with simple scoring system. Evaluations in two main areas: pain and sensorial exploration. The ﬁrst 5 questions asks for presence of unpleasant skin sensations (pricking, tingling, pins and needles), appearance of skin (mottled, red, or pink), increased sensitivity of skin to touch, sudden bursts of electric shock sensations, and hot or burning skin sensations. Last 2 questions involve sensory testing for the presence of allodynia and altered pinprick threshold. Different numbers of points, relative to their signiﬁcance to neuropathic pain, are given to positive answers for maximum of 24 points. A score less than 12 makes unlikely that participant's symptoms are neuropathic in nature, whereas score more than 12 make neuropathic mechanisms likely to be contributing to participant's pain. Change from baseline data has been calculated as value at baseline minus value at Day 84.
Time Frame: Baseline and Day 84 (Week 12)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Gabapentin/B-complex | Pregabalin
Number analyzed (Participants) | 147 | 123
units on a scale
  Baseline (n=147, 123) | 16.2 (3.6) | 15.8 (4.0)
  Change at Day 84 (n=146, 122) | 8.082 (7.470) | 6.967 (6.839)

3. Secondary Outcome: Change From Baseline in Visual Analogue Scale (VAS) Score at Day 84
Description: VAS is used to rate the pain as per 10 centimeter (cm) line. The pain intensity score ranges from '0=no pain' to '10=worst possible pain'. Change from baseline data has been calculated as value at baseline minus value at Day 84.
Time Frame: Baseline and Day 84 (Week 12)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: centimeter
Arm/Group | Gabapentin/B-complex | Pregabalin
Number analyzed (Participants) | 147 | 123
centimeter
  Baseline (n=147, 123) | 7.0 (1.8) | 7.1 (1.5)
  Change at Day 84 (n=146, 122) | 4.182 (2.890) | 4.529 (2.382)

4. Secondary Outcome: Profile of Mood States (POMS) Score
Description: POMS is a rating scale, which comprises of 65 items that are evaluated in a 0-4 scale, where 0 means "not at all" and 4 "extremely". The scores for the 65 items are added in various combinations to throw six validated factors which are used to calculate total POMS score: (tension-anxiety) + (depression-dejection) + (anger-hostility)+ (fatigue-Inertia) + (confusion-bewilderment) - (vigor-activity). Score range (-40 to 192). Score -40 denotes the best score and score 192 denotes the worst score.
Time Frame: Day 84 (Week 12)
Population: Per protocol population (PPP) included all the treated participants who showed no major protocol violations and were compliant with study inclusion criteria and with the proper administration of the study drug.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Gabapentin/B-complex | Pregabalin
Number analyzed (Participants) | 147 | 123
units on a scale | 1.3 (26.1) | 3.4 (25.5)

5. Secondary Outcome: Sleep Evaluation: Number of Participants Who Fell Asleep in Pre-specified Time Duration
Description: Sleep evaluation was performed by assessing number of participants who fell asleep in a particular pre-specified range of time duration, that is, 0-15 minutes, 16-30 minutes, 31-45 minutes, 46-60 minutes and greater than 60 minutes at Day 84 (Week 12).
Time Frame: Day 84 (Week 12)
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Gabapentin/B-complex | Pregabalin
Number analyzed (Participants) | 147 | 123
participants
  0 to 15 minutes | 85 (6.2) | 72 (5.4)
  16 to 30 minutes | 33 (2.8) | 33 (2.9)
  31 to 45 minutes | 13 | 12
  46 to 60 minutes | 8 | 4
  Greater than 60 minutes | 8 | 2

6. Secondary Outcome: Number of Participants With Various Health Conditions Based on Global Impression of Patient Change (GIPC) Scale
Description: GIPC is an assessment that the participant's global change in health condition from start of the study on a 7-point scale (1 = extremely improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse 6 = much worse, 7 = extremely worse).
Time Frame: Baseline and Day 84 (Week 12)
Population: Per protocol population (PPP) included all the treated participants who showed no major protocol violations and were compliant with study inclusion criteria and with the proper administration of the study drug. 'N' (number of participants analyzed) signifies participants who were evaluable for this measure.
Measure: Number; unit: participants
Arm/Group | Gabapentin/B-complex | Pregabalin
Number analyzed (Participants) | 145 | 122
participants
  Health: extremely improved | 62 | 47
  Health: much improved | 73 | 65
  Health: minimally improved | 10 | 10

7. Secondary Outcome: Number of Participants With Various Health Conditions Based on Clinical Global Impression of Change (CGIC) Scale
Description: CGIC is an assessment that the physician performs to assess the participant's global change in health condition from start of the study on a 7-point scale (1 = extremely improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse 6 = much worse, 7 = extremely worse).
Time Frame: Baseline and Day 84 (Week 12)
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | Gabapentin/B-complex | Pregabalin
Number analyzed (Participants) | 145 | 122
participants
  Health: extremely improved | 55 | 47
  Health: much improved | 79 | 69
  Health: minimally improved | 11 | 6

8. Secondary Outcome: Percentage of Participants With at Least 30 and 50 Percent (%) Improvement in Numeric Pain Intensity Scale (NPIS) From Baseline at Day 84 (Week 12)
Description: NPIS is a 11-point scale, with 0 representing no pain and 10 representing the worst possible pain. The participants were asked to mark the number that best represents the current level of pain they have experienced during the previous 24 hours.
Time Frame: Baseline and Day 84 (Week 12)
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Gabapentin/B-complex | Pregabalin
Number analyzed (Participants) | 147 | 123
percentage of participants
  At least 30% improvement | 76.9 | 85.4
  At least 50% improvement | 66.0 | 72.4

9. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An adverse event (AE) is defined as any untoward medical occurrence in the form of signs, symptoms, abnormal laboratory findings, or diseases that emerges or worsens relative to Baseline during a clinical study with an investigational medicinal product (IMP), regardless of causal relationship and even if no IMP has been administered.
Time Frame: Day 7 up to Day 84 (+7 days)
Population: Safety population included all the randomized participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Gabapentin/B-complex | Pregabalin
Number analyzed (Participants) | 174 | 174
participants | 80 | 93

ADVERSE EVENTS:
Time Frame: Day 7 up to Day 84 (+ 7 days)
Description: An AE is defined as any untoward medical occurrence in the form of signs, symptoms, abnormal laboratory findings, or diseases that emerges or worsens relative to Baseline during a clinical study with an IMP, regardless of causal relationship and even if no IMP has been administered.
Arm/Group | Gabapentin/B-complex | Pregabalin
Serious Adverse Events (participants affected / at risk) | 1/174 | 0/174
Other Adverse Events (participants affected / at risk) | 79/174 | 93/174
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gabapentin/B-complex (N=174) | Pregabalin (N=174)
Cerebrovascular disorder (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gabapentin/B-complex (N=174) | Pregabalin (N=174)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 2
Nervousness (Psychiatric disorders) | 0 | 1
Increased appetite (Metabolism and nutrition disorders) | 0 | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Asthenia (General disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 1
Cataract (Eye disorders) | 1 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Aphasia (Nervous system disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Prurigo (Skin and subcutaneous tissue disorders) | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 5 | 6
Insomnia (Psychiatric disorders) | 1 | 4
Movement disorder (Nervous system disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2 | 1
Flatulence (Gastrointestinal disorders) | 1 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 2
Constipation (Gastrointestinal disorders) | 1 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 14 | 13
Hypoacusis (Ear and labyrinth disorders) | 1 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 5
Vomiting (Gastrointestinal disorders) | 0 | 3
Dizziness (Nervous system disorders) | 32 | 52
Somnolence (Nervous system disorders) | 41 | 52
Vertigo (Ear and labyrinth disorders) | 1 | 11
Gait disturbance (General disorders) | 0 | 6
Fall (Injury, poisoning and procedural complications) | 0 | 1
Vascular insufficiency (Vascular disorders) | 1 | 0
Venous insufficiency (Vascular disorders) | 0 | 1
Eye irritation (Eye disorders) | 0 | 1
Oedema (Metabolism and nutrition disorders) | 2 | 3
Dry mouth (Gastrointestinal disorders) | 2 | 0
Odynophagia (Gastrointestinal disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 2 | 0
Intermittent claudication (Vascular disorders) | 0 | 1
Weight increased (Investigations) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1
Pityriasis (Skin and subcutaneous tissue disorders) | 1 | 0
Speech disorder (Nervous system disorders) | 0 | 1
Pharyngitis (Infections and infestations) | 2 | 2
Urinary tract infection (Infections and infestations) | 2 | 8
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
Vision blurred (Eye disorders) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No